CLINICAL TRIAL: NCT06831526
Title: A Window-of-opportunity Early Phase I Randomized Study of Neoadjuvant Chemoradiotherapy With or Without Concurrent Azeliragon in Patients With Newly Diagnosed Glioblastoma
Brief Title: Neoadjuvant Chemoradiotherapy With or Without Concurrent Azeliragon in Patients With Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cantex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202504190
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma
Keywords: GBM; Neoadjuvant chemoradiotherapy; Azeliragon; RAGE inhibitor; Window of opportunity study
MeSH Terms: conditions — Glioblastoma | interventions — azeliragon; Temozolomide; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Neoadjuvant RT and Temozolomide (TMZ) + Surgery or LITT + Adjuvant TMZ & Azeliragon (Active Comparator): Radiation therapy (RT) will consist of fractionated RT to 60 Gy in 30 daily fractions administered per standard of care RTOG approach. Concurrent TMZ during RT will be self-administered by mouth (PO) as per standard of care. 1 month after completion of RT, patient will proceed with planned surgery of either resection or LITT. Patients will then receive adjuvant TMZ and azeliragon for up to 6 months. Patient should start with the loading dose 30 mg BID for 6 days before the start of adjuvant TMZ. After 6 days, azeliragon 20 mg once daily should be continued in combination with TMZ.
  Interventions: Drug: Azeliragon; Drug: Temozolomide; Radiation: Radiation therapy; Procedure: Surgery or LITT
- Arm 2: Neoadjuvant RT, Temozolomide (TMZ) & Azeliragon + Surgery or LITT + Adjuvant TMZ & Azeliragon (Experimental): RT will consist of fractionated RT to 60 Gy in 30 daily fractions administered per standard of care RTOG approach. Concurrent TMZ during RT will be self-administered by mouth (PO) as per standard of care. Patients will receive azeliragon as well. Azeliragon is self-administered PO. Azeliragon dosing will consist of 6 days of a loading dose of 30 mg twice per day starting on day -6, followed by 20 mg daily starting on the Day 1. Concurrent RT and TMZ start on Day 1. Azeliragon should continue until the day before planned surgical procedure. 1 month after completion of RT, patient will proceed with planned surgery of either resection or LITT. Patients will then receive adjuvant TMZ and azeliragon for up to 6 months. Patient should start with the loading dose 30 mg BID for 6 days before the start of adjuvant TMZ. After 6 days, azeliragon 20 mg once daily should be continued in combination with TMZ.
  Interventions: Drug: Azeliragon; Drug: Temozolomide; Radiation: Radiation therapy; Procedure: Surgery or LITT

INTERVENTIONS:
Drug: Azeliragon — Provided by Cantex Pharmaceuticals
Drug: Temozolomide — Standard of care.
  Other Names: TMZ
Radiation: Radiation therapy — Standard of care.
Procedure: Surgery or LITT — Standard of care surgical resection or laser interstitial thermal therapy (LITT).

SUMMARY:
Preclinical data have demonstrated the combination of azeliragon, a RAGE inhibitor, with radiation therapy (RT) can effectively reduce immune-suppressive myeloid cells and restore T-cell activation to improve tumor control in murine glioma models. Ongoing clinical studies of azeliragon with RT alone and RT plus temozolomide (TMZ) to treat patients with newly diagnosed glioblastoma (GBM) have demonstrated safety and tolerability. The purpose of this window-of-opportunity study is to validate that the combination of azeliragon with RT and TMZ would modulate immune-suppressive myeloid and T cells in the tumor microenvironment in patients with GBM.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of IDH-wildtype GBM (WHO grade 4) according to the 2021 WHO classification (including subtypes such as gliosarcoma).
* Radiographic evidence of residual tumor after initial surgery or biopsy.
* Patient is amenable for future surgery (either surgical resection or laser interstitial thermal therapy (LITT)) to sample the residual tumor after completion of chemoradiotherapy.
* At least 18 years of age.
* Eligible for and planning to receive standard fractionated RT of 60 Gy with concurrent TMZ.
* Recovered from the effects of surgery, postoperative infection, and other complications sufficiently for initiation of chemoradiotherapy, in the opinion of the treating physician.
* Karnofsky performance status ≥ 60.
* Adequate organ and bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 K/cumm;
  * Platelets ≥ 100 K/cumm;
  * Hemoglobin > 9.0 g/dL (Note: the use of transfusion or other intervention to achieve Hgb >9.0 g/dL is acceptable);
  * Total bilirubin ≤ 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
  * Creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 mL/min
  * If there is history of human immunodeficiency virus (HIV) infection, patients must be on effective antiretroviral therapy, and HIV viral load must be undetectable within 6 months of study enrollment.
  * If there is history of chronic hepatitis B virus (HBV) infection, patients must have either been treated or are on suppressive therapy (as indicated), and HBV viral load must be undetectable.
  * If there is history of hepatitis C virus (HCV) infection, patients must have been treated, and HCV viral load must be undetectable.
* Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) and sexually active heterosexual males must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the trial and for 6 months after the last administration of azeliragon. Should a female trial participant or female partner of a male trial participants become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willingness to sign an IRB-approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior cranial RT or RT to the head and neck where potential field overlap may exist.
* Leptomeningeal or metastatic involvement.
* Known IDH mutation. IDH status could be determined by either immunohistochemistry or sequencing as evaluated per routine clinical care.
* Patients receiving CYP 2C8 inhibitors within 2 weeks or 5 half-lives prior to study entry.
* Patients with a gastrointestinal condition that could interfere with swallowing or absorption.
* Patients with concurrent participation in another interventional clinical trial or use of another investigational agent within 30 days prior to study entry. Patients who are participating in non-interventional clinical trials (e.g., QOL, imaging, observational, follow-up studies, etc.) are eligible, regardless of the timing of participation.
* Medical contraindication to MRI (e.g., unsafe foreign metallic implants, incompatible pacemaker, inability to lie still for long periods, severe to end-stage kidney disease or on hemodialysis).
* Pregnant or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of the first dose of RT (Arm 1) or azeliragon (Arm 2).
* Patients with psychiatric illness/social situations, including alcohol or drug abuse that in the investigator's opinion will prevent administration or completion of protocol therapy.
* Non-English speaking, as the cognitive assessments will only be available in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of immune-suppressive myeloid cells in the tumor tissue | At time of surgery or LITT (estimated to be day 60)
Percentage of immune-suppressive T cells in the tumor tissue | At time of surgery or LITT (estimated to be day 60)

SECONDARY OUTCOMES:
Number of participants with adverse events | From day 1 (Arm 1) or Day -6 (Arm 2) through 30 days after last dose of azeliragon (estimated to be 10 months)
Number of participants with intolerable toxicities | From first dose of azeliragon until 30 days after the last dose (estimated to be 6-9 months)
  The protocol lists the specific toxicities that are considered intolerable.
Progression-free survival (PFS) | Up to 12 months after completion of study treatment (estimated to be 21 months)
Overall survival (OS) | Up to 12 months after completion of study treatment (estimated to be 21 months)
Feasibility of the regimen as measured by the number of participants who proceed with post-chemoradiotherapy surgery or LITT | Through surgery or LITT (estimated to be 60 days)
  Feasibility is defined as at least 50% of patients in each arm who are able to proceed with post-chemoradiotherapy surgery or LITT.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu